CLINICAL TRIAL: NCT04621461
Title: A Randomized, Placebo-Controlled Study Evaluating the Efficacy of Zinc for the Treatment of COVID-19 in the Outpatient Setting
Brief Title: Placebo Controlled Trial to Evaluate Zinc for the Treatment of COVID-19 in the Outpatient Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20-19
Record Dates: First submitted 2020-11-06; First posted 2020-11-09 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Corona Virus Infection
Keywords: COVID-19; Zinc
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Zinc Sulfate

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled trial to assess the efficacy of zinc in a higher risk COVID-19 positive outpatient population. Patients will randomized to zinc or placebo.
Who Masked: Participant, Investigator
Masking Description: Patients will be randomized via a randomization block. Only the research coordinator will know which group the patients belong to. Placebo pills given to the patient will be similar in size and shape to zinc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm #1 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Experimental Arm #2 (Experimental): Zinc sulfate
  Interventions: Dietary Supplement: Zinc Sulfate 220 MG

INTERVENTIONS:
Dietary Supplement: Zinc Sulfate 220 MG — 220mg once daily for 5 days
  Arms: Experimental Arm #2
Drug: Placebo — Once daily for 5 days
  Arms: Experimental Arm #1

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial to assess the efficacy of zinc in a higher risk COVID-19 positive outpatient population.

DETAILED DESCRIPTION:
Zinc, a micronutrient, appears to have anti-viral properties with various mechanisms of action depending on the concentration Zinc supplementation has been reviewed extensively for use in the common cold, and has been shown to reduce the duration of symptoms. In-vitro studies have shown zinc can inhibit RNA-dependent RNA polymerase (RdRP) in coronavirus, which is typically a conserved region in the viral genome. In-vitro experiments have also shown that lung epithelium in a zinc depleted state can become susceptible to apoptosis and loss of barrier function, increasing permeability, which can lead to acute respiratory distress syndrome (ARDS).

If a patient can travel to St. Francis Hospital they can have a COVID test on site at a designated St. Francis testing location. The COVID test will be resulted via a rapid Covid (Point of Care device) or at a local lab.

Patients who are unable to travel to St. Francis Hospital or one of the outpatient practices, will be allowed to enroll remotely. Patients are eligible to enroll within 72 hours of a positive Covid-19 test result. Study medications will be mailed to the patient overnight after being enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand informed consent.
* High initial clinical suspicion by physician based on signs and symptoms (fever, cough, myalgias, fatigue, shortness of breath) followed by confirmation of COVID-19 diagnosis
* Any gender
* Age 60 years and older
* Age 30-59 years with one or more of the following:

  * abnormal lung exam
  * abnormal oxygen saturation <95%
  * abnormal Chest X-ray or chest CT
  * persistent fever >100.4 degrees Fahrenheit
  * one of the following co-morbidities: hypertension, diabetes mellitus, history of coronary artery disease, chronic kidney disease (CKD), asthma, COPD, current or former smoker, or morbid obesity (Body Mass Index ≥35)

Exclusion Criteria:

* Severe COVID-19 requiring admission for inpatient treatment
* Need for any oxygen supplementation
* Need for mechanical ventilatory support
* History of oxygen supplementation dependency
* History of cancer with ongoing chemotherapy or radiation therapy
* Known hypersensitivity to zinc
* Severe renal disease: Glomerular Filtration Rate <30ml/min

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Number of participants hospitalized and/or requiring repeat emergency room visits | 21 days
  COVID-19 related complications that require the participant to be hospitalized or have an emergency room visit
Number of participants admitted to the Intensive care unit (ICU) | 30 days
  If hospitalized, number of participants admitted to the ICU, and number of days in the ICU
Number of participants on a ventilator | 30 days
  If placed on ventilator, number of days on a ventilator

SECONDARY OUTCOMES:
All-cause mortality | Up to 30 days
  Total number of deaths in the cohort.
Time to resolution of COVID-19 symptoms | Evaluated at day 2, 6, day 14, and day 21
  Time at which the patient is completely symptom free.
Severity of symptoms | Evaluated at day 2, 6, day 14, and day 21
  Scored by the participant for feverishness, sore throat, cough, shortness of breath, myalgias. (0 =none; 1 = mild; 2 = moderate; 3 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Avni Thakore, MD, Principal Investigator — St. Francis Hospital - The Heart Center
Locations (1):
- St. Francis Hospital - The Heart Center, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu C, Liu Y, Yang Y, Zhang P, Zhong W, Wang Y, Wang Q, Xu Y, Li M, Li X, Zheng M, Chen L, Li H. Analysis of therapeutic targets for SARS-CoV-2 and discovery of potential drugs by computational methods. Acta Pharm Sin B. 2020 May;10(5):766-788. doi: 10.1016/j.apsb.2020.02.008. Epub 2020 Feb 27. PMID 32292689
- [Background] Korant BD, Butterworth BE. Inhibition by zinc of rhinovirus protein cleavage: interaction of zinc with capsid polypeptides. J Virol. 1976 Apr;18(1):298-306. doi: 10.1128/JVI.18.1.298-306.1976. PMID 176466
- [Background] Katz E, Margalith E. Inhibition of vaccinia virus maturation by zinc chloride. Antimicrob Agents Chemother. 1981 Feb;19(2):213-7. doi: 10.1128/AAC.19.2.213. PMID 7347557
- [Background] Kumel G, Schrader S, Zentgraf H, Daus H, Brendel M. The mechanism of the antiherpetic activity of zinc sulphate. J Gen Virol. 1990 Dec;71 ( Pt 12):2989-97. doi: 10.1099/0022-1317-71-12-2989. PMID 2177090
- [Background] Suara RO, Crowe JE Jr. Effect of zinc salts on respiratory syncytial virus replication. Antimicrob Agents Chemother. 2004 Mar;48(3):783-90. doi: 10.1128/AAC.48.3.783-790.2004. PMID 14982765
- [Background] Eby GA, Davis DR, Halcomb WW. Reduction in duration of common colds by zinc gluconate lozenges in a double-blind study. Antimicrob Agents Chemother. 1984 Jan;25(1):20-4. doi: 10.1128/AAC.25.1.20. PMID 6367635
- [Background] te Velthuis AJ, van den Worm SH, Sims AC, Baric RS, Snijder EJ, van Hemert MJ. Zn(2+) inhibits coronavirus and arterivirus RNA polymerase activity in vitro and zinc ionophores block the replication of these viruses in cell culture. PLoS Pathog. 2010 Nov 4;6(11):e1001176. doi: 10.1371/journal.ppat.1001176. PMID 21079686
- [Background] Singh M, Das RR. Zinc for the common cold. Cochrane Database Syst Rev. 2013 Jun 18;(6):CD001364. doi: 10.1002/14651858.CD001364.pub4. PMID 23775705
- [Background] Bao S, Knoell DL. Zinc modulates airway epithelium susceptibility to death receptor-mediated apoptosis. Am J Physiol Lung Cell Mol Physiol. 2006 Mar;290(3):L433-41. doi: 10.1152/ajplung.00341.2005. Epub 2005 Nov 11. PMID 16284213